CLINICAL TRIAL: NCT00491426
Title: Antimicrobial Pharmacokinetics in High Risk Infants (Urinary Proteomics in Antimicrobial/Antifungal-Treated Newborns - add-on Study)
Brief Title: Antimicrobial PK in Infants With Suspected or Confirmed Infection
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Pediatric Pharmacology Research Units Network (Network)
Responsible Party: Sponsor
Other Study IDs: Pro00015379; PPRU 10824 (Other: Network Protocol Identifier)
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Infection
Keywords: Infection; Anti-Infective Agents; Antifungal Agents; Proteomics
MeSH Terms: conditions — Infections | interventions — Ampicillin; Metronidazole; Piperacillin, Tazobactam Drug Combination; Acyclovir; Amphotericin B; liposomal amphotericin B; Anidulafungin; Caspofungin

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- <26 weeks: Subjects <26 weeks gestational age
  Interventions: Drug: Ampicillin; Drug: Metronidazole; Drug: Piperacillin/Tazobactam; Drug: Acyclovir; Drug: Amphotericin B; Drug: Ambisome; Drug: Anidulafungin; Drug: Caspofungin
- 26-29 weeks: Subjects 26-29 weeks gestational age
  Interventions: Drug: Ampicillin; Drug: Metronidazole; Drug: Piperacillin/Tazobactam; Drug: Acyclovir; Drug: Amphotericin B; Drug: Ambisome; Drug: Anidulafungin; Drug: Caspofungin
- 30-32 weeks: Subjects 30-32 weeks gestational age
  Interventions: Drug: Ampicillin; Drug: Metronidazole; Drug: Piperacillin/Tazobactam; Drug: Acyclovir; Drug: Amphotericin B; Drug: Ambisome; Drug: Anidulafungin; Drug: Caspofungin

INTERVENTIONS:
Drug: Ampicillin — Drug prescribed per routine medical care.
Drug: Metronidazole — Drug prescribed per routine medical care.
Drug: Piperacillin/Tazobactam — Drug prescribed per routine medical care.
Drug: Acyclovir — Drug prescribed per routine medical care.
Drug: Amphotericin B — Drug prescribed per routine medical care.
Drug: Ambisome — Drug prescribed per routine medical care.
Drug: Anidulafungin — Drug prescribed per routine medical care.
Drug: Caspofungin — Drug prescribed per routine medical care.

SUMMARY:
The purpose of this protocol is to provide a mechanism for the ongoing collection of blood and urine samples in newborns that will be used to measure levels of antimicrobial products used in the newborn population where there are limited pharmacokinetic data in either premature or term infants.

DETAILED DESCRIPTION:
Greater than 90% of infants born <32 weeks admitted to critical care nurseries are treated with antimicrobial agents during their NICU hospitalization. Most antimicrobial products used in the neonatal population lack some aspect of pharmacokinetic information specific to neonates. Dosing is based largely on pharmacokinetic data from older children or in some cases, adults. This study will also establish a bank of urine samples from newborns treated with antimicrobial and/or antifungal therapy and to characterize the urinary proteome in selected samples. The sites of the NIH-sponsored Pediatric Pharmacology Research Network (PPRU) have access to appropriate assays using microliter amounts of serum and a large pool of potential subjects to generate meaningful data that will

1. Guide dosing of commonly used antimicrobial agents, and
2. Provide preliminary data for future industry and government trials in the nursery.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≤32 weeks and 6 days EGA with high probability of receiving one of the antimicrobial agents listed are eligible for study.
* Age younger than 120 days
* Written informed consent from parent or legal guardian
* Infants likely to survive beyond 48 hours after enrollment

Exclusion Criteria:

* Failure to consent

Max Age: 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants <32 weeks gestational age at birth at risk of infections.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2006-01; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Benjamin, MD, Principal Investigator — PPRU; Mary Jayne Kennedy, Pharm, D, Principal Investigator — Louisville-PPRU
Locations (6):
- United States (6):
  - University of California at San Diego, La Jolla, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital of Michigan, Wayne State University, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas